CLINICAL TRIAL: NCT01824914
Title: Comparison of Cormack-Lehane Score in Sedation and Anesthesia Condition by McGrath Videolaryngoscope
Brief Title: Airway Evaluation by McGrath Videolaryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wenlong Yao, M.D., Ph.D., Attending physician, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: TJMZK20121231
Record Dates: First submitted 2013-03-25; First posted 2013-04-05 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Anesthesia
Keywords: videolaryngoscope; tracheal intubation; Cormack-Lehane grade; airway evaluation; sedation; anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- McGrath Videolaryngoscope (Experimental): to compare the Cormack-Lehane grade in sedation and anesthesia by McGrath videolaryngoscope
  Interventions: Device: McGrath Videolaryngoscope

INTERVENTIONS:
Device: McGrath Videolaryngoscope — A kind of portable videolaryngoscopes, produced by Aircraft Medical. It has been used for difficult airway.

SUMMARY:
Difficult tracheal intubation is a cause of severe patient damage and death. There is not a good method to predict it. The McGrath Series 5 video laryngoscope can improve visualization of the glottic structures one to two grades. Moreover unlike a classical laryngoscope with a Macintosh blade, the McGrath provides a view of the glottis without requiring alignment of the oral, pharyngeal and laryngeal axes. In this study, the investigators will use it to compare the Cormack-Lehane score in sedation and anesthesia condition. It helps to know the role of videolaryngoscope in predicting difficult intubation.

DETAILED DESCRIPTION:
* The enrolled patients were given a bolus of sufentanil 0.3-0.5μg/kg to achieve Ramsay sedation score 2-3. The Cormack-Lehane score in sedation was evaluated by McGrath videolaryngoscope.
* Then the patients were induced with propofol. A bolus of rocuronium was given to facilitate intubation. The Cormack-Lehane score in anesthesia was recorded when intubated by McGrath videolaryngoscope.
* BMI, mouth opening, thyromental distance, intubation duration and ramsay sedation score were also recorded.
* To compare the Cormack-Lehane score in sedate and anesthesia condition

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for general surgery under general anesthesia
* ASA classification 1-3

Exclusion Criteria:

* emergent operation, aspiration risk
* a history of difficult airway
* expected difficult airway
* incooperative patients with mental diseases, hearing disorders

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Cormack-Lehane score in sedation condition | 5 minutes after administration of sufentanil
  Based on the Modified Cormack-Lehane classification. 5 degrades. 1-5
Cormack-lehane score in anesthesia condition | 1 minute after administration of rocuronium
  Based on the Modified Cormack-Lehane classification. 5 degrades. 1-5

SECONDARY OUTCOMES:
Duration of intubation | At intubation
  The duration of intubation is defined as the time from inserting videolaryngoscope, intubating a tube, to withdrawing videolaryngoscope using a stopwatch.
Sedation score | 5 minutes after administraion of sufentanil
  by Ramsay sedation score 1-6. The higher score, the deeper sedation

OTHER OUTCOMES:
BMI | One day before operation
Thyromental distance | One day before operation
  measuring with a ruler
Mallampati classification | One day before operation
  4 degrades
Mouth opening | One day before operation
  measuring with a ruler

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, Ph.D.,M.D., Study Director — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China